CLINICAL TRIAL: NCT05659381
Title: GOG-3068: A Phase III Randomized Trial of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) With Cisplatin Versus no HIPEC at the Time of Optimal Interval Cytoreductive Surgery Followed by Niraparib Maintenance in Patients With Homologous Recombinant Deficient (HRD +) Newly Diagnosed Stage III and IV Ovarian, Primary Peritoneal, and Fallopian Tube Cancer (Heated Ovarian Treatment Trial)
Brief Title: Heated Intraperitoneal Chemotherapy Followed by Niraparib for Ovarian, Primary Peritoneal and Fallopian Tube Cancer
Acronym: HOTT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3068; 217908 (Other: GSK)
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Stage III Primary Peritoneal Cancer; Stage IV Primary Peritoneal Cancer; Stage III Fallopian Tube Cancer; Stage IV Fallopian Tube Cancer
Keywords: HIPEC
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIPEC (Experimental): Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Cisplatin 100 mg/m2 IP over 90 minutes at 42 degrees C
  Interventions: Drug: Cisplatin
- No HIPEC (Active Comparator): No treatment
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 100mg/m2 IP over 90 minutes at 42 degrees Celcius
  Other Names: Platinol AQ
  Arms: HIPEC
Other: No treatment — No treatment with Cisplatin
  Arms: No HIPEC

SUMMARY:
Patients will be registered prior to, during or at the completion of neoadjuvant chemotherapy given per standard institutional guidelines +/- bevacizumab on Day 1 every 21 days for 3-4 cycles. Registered patients who progress during neoadjuvant chemotherapy will not be eligible for iCRS and will be removed from the study.

Following completion of neoadjuvant chemotherapy, interval cytoreductive surgery (iCRS) will be performed in the usual fashion in both arms. Patients will be randomized at the time of iCRS (iCRS must achieve no gross residual disease or no disease >1.0 cm in largest diameter) to receive HIPEC or no HIPEC. Patients randomized to HIPEC Arm will receive a single dose of cisplatin (100mg/m2 IP over 90 minutes at 42 C) as HIPEC. After postoperative recovery patients will receive standard post-operative platinum-based combination chemotherapy. Patients randomized to surgery only (No HIPEC Arm) will receive postoperative standard chemotherapy after recovery from surgery.

Both groups will receive an additional 2-3 cycles of platinum-based combination chemotherapy per standard institutional guidelines +/- bevacizumab for a maximum total of 6 cycles of chemotherapy (neoadjuvant plus post-operative cycles) followed by niraparib individualized dosing +/- bevacizumab until progression or 36 months (if no evidence of disease).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a pathologic diagnosis of high grade serous or endometroid epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, FIGO stage III or IV documented on CT scan/MRI, must be recommended and agree to undergo platinum-based neoadjuvant chemotherapy with or without physician choice bevacizumab (3-4 cycles allowed, with bevacizumab held for at least 28 days preoperatively) and are considered candidates for (and planned to have) interval cytoreductive surgery (iCRS) followed by chemotherapy and niraparib maintenance as determined by the enrolling investigator. Patients may continue bevacizumab after a minimum of 28 days post iCRS and during niraparib maintenance per local standard.
2. Patients with stage IV disease must have complete response of extra-abdominal disease on preoperative imaging (e.g. pleural effusion, mediastinal, inguinal, supraclavicular lymphadenopathy, or other extra-abdominal metastases) or be deemed resectable with iCRS.
3. Patients must have HRD/LOH positive tumors. Patients with germline or somatic BRCA or other similar mutations (RAD51C, RAD51D, BRIP1, BARD) are not required to have HRD/LOH testing. Patients without BRCA or germline mutations must have HRD/LOH testing using Myriad myChoice®/Foundation Medicine/Caris Life Sciences platforms. HRD test results must be available prior to registration to meet entry criteria.
4. Patients must have R0 (no gross/visible residual disease) or R1 (gross/visible residual disease ≤ 1.0 cm in the longest diameter) following iCRS and prior to randomization.
5. Patient must have adequate bone marrow and organ function:

   Bone marrow function:

   Hemoglobin ≥ 8.5 g/dL. Absolute neutrophil count (ANC) ≥ 1,500/mm3. Platelets ≥ 100,000/mm3.

   Renal function:

   Creatinine ≤ 1.3mg/dl OR Calculated creatinine clearance (≥ 30 mL/min/1.73 m2) per National Kidney Foundation guidelines and NHANES III

   Hepatic function:

   Bilirubin ≤ 1.5 times ULN. ALT ≤ 3 times the ULN. AST ≤ 3 times the ULN.

   Neurologic function:

   Peripheral neuropathy ≤ CTC AE grade 2.
6. Patients must have an ECOG performance status of 0 or 1.
7. Patient must be age > 18.
8. Patients must have a life expectancy > 3 months.
9. Patients of childbearing potential must have a negative serum pregnancy test within 28 days prior to iCRS and must be practicing an effective form of contraception (with failure rate <1% per year) during the study period and for 6 months following the last dose of niraparib. Patients of childbearing potential must consent to pregnancy testing prior to receiving niraparib and monthly thereafter for the duration of the study.

   Patients are considered postmenopausal and not of child-bearing potential if they are free from menses for >1 year or surgically sterilized.
10. Patients must have normal blood pressure (BP) or adequately treated and controlled hypertension based on local standard of care (systolic BP ≤ 140 mmHg and diastolic ≤ 90 mmHg) prior to starting niraparib.
11. Patients receiving corticosteroids may continue as long as their dose is stable for at least 4 weeks prior to randomization.
12. Patients must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
13. Patients with known human immunodeficiency virus (HIV) are allowed if they meet all the following criteria:

    1. Cluster of differentiation 4 ≥350/µL and viral load <400 copies/mL
    2. No history of acquired immunodeficiency syndrome-defining opportunistic infections within 12 months prior to enrollment
    3. No history of HIV associated malignancy for the past 5 years
    4. Concurrent antiretroviral therapy as per the most current National Institutes of Health (NIH) Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV started >4 weeks prior to study enrollment
14. Patient or a legally authorized representative must have signed an approved informed consent and authorization permitting the release of personal health information.

Exclusion Criteria

1. Patients with low-grade serous, clear cell, mucinous, non-epithelial ovarian cancers and borderline tumors.
2. Patients who have received prior treatment for ovarian cancer other than the first 3-4 cycles of platinum based neoadjuvant chemotherapy. Prior neoadjuvant treatment with bevacizumab is allowed; bevacizumab must be held for 28 days prior to surgery.
3. Patients whose tumors are HRD/LOH negative.
4. Patients not eligible for iCRS based on evidence of progression of disease during neoadjuvant chemotherapy (documented on CT scan/MRI required within 35 days of iCRS).
5. Patients not eligible for iCRS based on medical co-morbidities as per the enrolling investigator.
6. Patients with stage IV disease without complete response of extra-abdominal disease on preoperative findings (e.g., pleural effusion, mediastinal, inguinal, supraclavicular lymphadenopathy, mesemchymal liver metastases or other extra-abdominal metastases) who are not deemed resectable with iCRS.
7. Patients with a history of Myelodysplastic Syndrome or Acute Myeloid Leukemia.
8. Patients who are pregnant or lactating.
9. Patients with a severe infection requiring IV antibiotics within 2 weeks of planned randomization.
10. Patients with other uncontrolled, intercurrent medical conditions.
11. Patient with metastatic disease to the central nervous system.
12. Patient with uncontrolled insulin dependent diabetes or pre-existing renal condition.
13. Patients with pre-existing hearing loss related to prior platinum-based chemotherapy.
14. Patients with Prior Reversible Encephalopathy Syndrome (PRES).
15. Patients with current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment). Severe hepatic impairment patients should be excluded.
16. Patients with any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels that is not related to ovarian cancer.
17. Patients with clinically significant cardiovascular disease (e.g., significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, uncontrolled cardiac arrhythmia or unstable angina <6 months to randomization, New York Heart Association Grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade 2 or greater peripheral vascular disease, and history of cerebrovascular accident within 6 months).
18. Patients with an increased bleeding risk due to concurrent conditions (e.g., major injuries or major surgery within the past 28 days prior to study randomization and/or history of hemorrhagic stroke, transient ischemic attack, subarachnoid hemorrhage, or clinically significant hemorrhage within the past 3 months).
19. Patients with known active hepatitis B (eg, hepatitis B surface antigen reactive) are excluded unless their HBV is stably controlled on nucleos(t)ide analogs (eg entecavir or tenofovir) which will be continued for the duration of the study.
20. Patient has had investigational therapy administered within 4 weeks or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to study randomization.
21. Patient has received a live vaccine within 30 days of study randomization. COVID-19 vaccines that do not contain live viruses are allowed at any time during the study.
22. Patient has a diagnosis, detection, or treatment of another type of invasive cancer ≤ 2 years prior to initiating protocol therapy (except for basal or squamous cell carcinoma of the skin, cervical cancer in situ, and ductal cancer in situ (DCIS) that has been definitively treated).
23. Patients must not have had radiotherapy encompassing > 20% of the bone marrow within 2 weeks of randomization; or any radiation therapy within 1 week prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 220 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2034-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From enrollment until time of disease progression or death, whichever occurs first, or date of last contact if neither progression of death has occurred, assessed up to 8 years
  Progression free survival in patients who receive a single treatment of intraoperative HIPEC with cisplatin vs. those who do not receive intraoperative HIPEC with cisplatin.

SECONDARY OUTCOMES:
Overall Survival | From enrollment to the time of death or date of last contact, assessed up to 8 years
  Overall survival stratified by:
  1. Stage at diagnosis (stage III vs. stage IV)
  2. Germline or somatic mutation (yes vs. no)
  3. Physician choice bevacizumab (yes vs. no)
  4. Residual disease (no gross/visible residual disease vs. gross/visible residual disease less than or equal to 1 cm in longest diameter
Frequency and severity of adverse events | Every 28 days up to 3 years
  The frequency and severity of adverse events as defined by CTCAE version 5.0
Progression Free Survival | From the time of randomization until the date of first documented disease progression or death from any cause, whichever came first, assessed up to 8 years
  Progression Free Survival stratified by:
  1. Stage at diagnosis (stage III vs. stage IV)
  2. Germline or somatic mutation (yes vs. no)
  3. Physician choice bevacizumab (yes vs. no)
  4. Residual disease (no gross/visible residual disease vs. gross/visible residual disease less than or equal to 1 cm in longest diameter

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Randall, MD, Study Chair — GOG Foundation
Locations (58):
- United States (58):
  - City of Hope, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Ambulatory Surgery Center Lane Operating Room, Palo Alto, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Stanford Hospital, Palo Alto, California
  - University of Colorado Hospital - Anshutz Cancer Pavilion, Aurora, Colorado
  - Smilow Cancer Hospital at Yale- New Haven, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Sylvester Comprehensive Cancer Center - The Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami Hospital and Clinics - Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Sylvester Comprehensive Cancer Center - Plantation, Plantation, Florida
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Medical Center MOB, Kansas City, Kansas
  - University of Kansas Cancer Center Overland Park, Overland Park, Kansas
  - University of Kansas Indian Creek Breast Surgery, Overland Park, Kansas
  - University of Kansas Cancer Center Westwood, Westwood, Kansas
  - University of Kansas Clinical Research Center, Westwood, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - LSU Health New Orleans, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - University of Kansas Cancer Center, Kansas City, Missouri
  - University of Kansas Cancer Center North, Kansas City, Missouri
  - University of Kansas Cancer Center Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - UH Geauga Medical Center, Chardon, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - TriHealth Cancer Institute - Good Samaritan Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute- Thomas Comprehensive Care Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - SCC at Lake University, Mentor, Ohio
  - UH Minoff Health Center at Chagrin Highlands, Orange, Ohio
  - West Chester Hospital, West Chester, Ohio
  - St. John Medical Center, Westlake, Ohio
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Wexford Hospital, Wexford, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center/Mainline Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina (Hollings Cancer Center), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Central South, Austin, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - O'Quinn Medical Tower at McNair Campus, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Froedtert Memorial Lutheran Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin